CLINICAL TRIAL: NCT04336046
Title: Ultrasound Guided Bilateral Erector Spinae Block as Analgesia for Adolescent Idiopathic Scoliosis Correction
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: busy
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Faheem, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: bilateral erector spinae block
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Erector Spinae Block; Analgesia; Scoliosis Idiopathic
MeSH Terms: conditions — Agnosia | interventions — Saline Solution; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Sham Comparator): will receive sham bilateral ultrasounded guided erector spinae block using 1 mg /kg normal saline in a total volume of 20 ml for each side after induction of anaesthesia in prone position after induction of anaesthesia in prone position.
  Interventions: Procedure: sham bilateral ultrasounded guided erector spinae block; Drug: normal saline
- erector spinae block (Experimental): will receive real bilateral ultrasounded guided erector spinae block by bupivacaine at 1 mg /kg in a total volume of 20 ml for each side after induction of anaesthesia in prone position
  Interventions: Procedure: erector spinae block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: erector spinae block — will receive real bilateral ultrasounded guided erector spinae block by bupivacaine at 1 mg /kg in a total volume of 20 ml for each side after induction of anaesthesia in prone position
  Arms: erector spinae block
Procedure: sham bilateral ultrasounded guided erector spinae block — will receive sham bilateral ultrasounded guided erector spinae block using 1 mg /kg normal saline in a total volume of 20 ml for each side after induction of anaesthesia in prone position after induction of anaesthesia in prone position.
  Arms: control group
Drug: normal saline — using 1 mg /kg normal saline
  Arms: control group
Drug: Bupivacaine — bupivacaine
  Arms: erector spinae block

SUMMARY:
Scoliosis is a structural, tridimensional deformity of the spine. Characterized by lateral curvature and rotation of the vertebrae with functional limitations and cosmetic problems, idiopathic scoliosis, which accounts for 75% to 80% of all scoliosis, is the most common of all types. (1, 2) Surgical treatment is an effective way to correct severe spine deformity when the deformity progressively worsens and cannot be positively corrected by brace treatment. Spinal correction surgery is one of the most invasive surgical procedures and usually results in moderate to severe levels of postoperative pain. (3) Severe pain may induce implant complications such as construct dislodgement, broken instrumentation, and implant loosening which requires additional revision procedures These conditions adversely affect postoperative outcomes.(4) In the past several years, pain has become an important indicator for evaluating indicators of outcome and quality of life after surgery. Effective analgesia after surgery could improve patients' prognosis.(5) The erector spinae block is a recently described ultrasound-guided technique in which local anesthetics is injected into a fascial plane between the tips of the thoracic transverse processes and the overlying erector spinae muscle (longissimus thoracis).(6) The available evidence indicates that erector spinae block is effective in reducing opioid requirements and improving the pain experience in a wide range of clinical settings. They are best employed as part of multimodal analgesia with other systemic analgesics

DETAILED DESCRIPTION:
-Preoperative: Evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigation and patients will be trained to use the Numerical Rating Scale (NRS 0= no pain, 10= intolerable pain) used for evaluation of pain intensity.

The patient is allowed to fast for 8 hours for solids and 2h for clear fluid. Before the study, all patients will be interviewed and will be briefed on the wake-up test procedure. They will be informed that they will be asked to open their eyes, move their fingers (hold the anesthesiologist's hand), move their toes, and finally, to remember a given color.

-Intraoperative: On arrival to operating roome, a 20 G peripheral IV cannula will be inserted. Electrocardiogram (ECG), noninvasive mean arterial blood pressure (MAP) and peripheral oxygen saturation will be attached and baseline data will be monitored and documented. Sedation will be given intravenously in the form of midazolam 0.02 mg/kg and IV fliud according to calculation of deficit and maintaince calculation.

After preoxygenation, anesthesia with IV propofol 2 mg/ kg and fentanyl 2 µg/kg will be administered for analgesia and cisatracurium 0.5 mg/ kg will be given intravenously to facilitate endotracheal intubation.

Central venous catheter will be inserted and attached for monitoring of CVP. Also, enotropy will be connected on the patientꞌs forehead and maintained between 40-60.

40 patients will be equally divided to two equal groups (20 patients for each group) Group 1: will receive sham bilateral ultrasounded guided erector spinae block using 1 mg /kg normal saline in a total volume of 20 ml for each side after induction of anaesthesia in prone position after induction of anaesthesia in prone position.

Group 2: will receive real bilateral ultrasounded guided erector spinae block by bupivacaine at 1 mg /kg in a total volume of 20 ml for each side after induction of anaesthesia in prone position.

Maintaince of anaesthesia will be 50 : 50 % O2 to air and sevoflurane 2% and cisatracurium incremental every 30 min at dose of 0.1 mg/kg. I.V analgesia in form of incremental fentanyl 1 ug /kg when entropy increases more than 60 during surgery and 30 min before the wake-up test.

Wake up test: Before continuation of anesthesia, patients will be given a color to remember. After finishing the wake-up test, anesthesia will be induced using 3 mg/kg propofol and 0.1 mg/kg cisatracurium, whereas anesthesia will be maintained as described previously.

At the end of surgery, inhalational anesthetic agent will be turned off, residual neuromuscular block will be reversed with neostigmine 0.05 mg/kg and atropine 0.01 mg/kg then patients will be extubated and will be transferred to post anesthesia care unit (PACU).

Postoperative multimodal analgesia: will received paracetamol 10 mg/kg every 6 hours and intravenous diclofenac 1.5 mg/kg every 8 hours regularly.

All observations will be carried out by a single investigator, who is blinded to the study groups.

-In all groups, the following will be measured: -

1. Demographic data.
2. Total doses of postoperative morphine consumption.
3. Time of the first dose of rescue analgesia (morphine at dose of 0.1 mg/kg).
4. Number of patients received rescue analgesia.
5. Numerical Rating Scale (NRS) for pain that ranged from (0 = no pain) to (10 = intolerable pain). If score is >3 will need analgesia in the form of morphine 0.1 mg/kg will be given till NRS decreases to ≤3. NRS will be assessed and recorded on arrival to the Recovery Unit, 2, 4, 8, 12, 18, 24 h after the operation, by an anesthesiologist, who is blinded to the study groups.
6. Total doses intraoperative consumption of fentanyl.
7. Wake-up profile: On the surgeons' request for the intraoperative wake-up test, administration of sevoflurane will be stopped. (the quality of wake-up, return of spontaneous breathing, ability to open eyes on command, and ability to move hands and feet) and postoperative amnesia. Patients will be asked repeatedly during the wake-up test, at least every 15 s, to open their eyes and to move their hands and feet. The time elapsed from the interruption of anesthesia to the start of spontaneous breathing (T1), from the return of spontaneous breathing to eye opening on command (T2), and from eye opening to movement of hands and feet (T3) will be recorded in seconds using a stopwatch. The quality of the wake-up test will be evaluated on a three-point rank scale (8).
8. First time of postoperative mobilization.

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopathic adolescent scoliosis undergoing surgical correction.

Exclusion Criteria:

* Bleeding disorders (coagulopathy).
* Mental dysfunction.
* History of allergy to local anesthetics.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
postoperative morphine consumption | within 24 hours postoperative
  postoperative morphine consumption

SECONDARY OUTCOMES:
intraoperative fentanyl consumption | intraoperative
  intraoperative fentanyl consumption
time to first analgesic request | within 24 hours postoperative
  time to first analgesic request

CONTACTS AND LOCATIONS:
Locations (1):
- tarek Abdel Lattif, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No